CLINICAL TRIAL: NCT02891889
Title: Description of the Appearance of Brown Fat in Scanner
Acronym: BAT
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: BAT
Record Dates: First submitted 2016-08-30; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Description of Brown Fat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to investigate aspects of brown fat in scanner with injection via the PET-CT study.

DETAILED DESCRIPTION:
Brown fat is metabolically active adipose tissue. It can be responsible in PET-CT of a fixation of 18-FDG and a look of pseudo-infiltration of fat. These aspects can be sources of false positives. The objective here is to gain a better knowledge of the scanner in areas of brown fat.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients since June 2014, who underwent a thoraco-abdominopelvic PET-CT examination with 18F-FDG in the University Hospital of Brest, in a clinical setting which warranted.
* Major Patients
* No opposition formalized

Exclusion Criteria:

* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients had a thoraco-abdominopelvic PET-CT examination with18F-FDG in a clinical setting which warranted.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Density value | 1 year
  measured by CT and expressed in Hounsfield Units

SECONDARY OUTCOMES:
Standard Uptake Values (SUV) adipose tissue "white" and "brown". | 1 year
  SUV maximum and average

CONTACTS AND LOCATIONS:
Overall Officials: Douraied Ben Salem, Professor, Principal Investigator — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France